CLINICAL TRIAL: NCT03116464
Title: Family Telemental Health Intervention for Veterans With Dementia
Acronym: TMH Pilot
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment and resources to continue the study
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPO 16-131; I21HX002256 (NIH)
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Dementia Family Caregiver Burden and Conflict

STUDY DESIGN:
Intervention Model Description: Family based telemental health intervention that incorporates: (1) psychoeducation on dementia, (2) communication and problem solving skills, (3) safety building skills, (4) relationship satisfaction enhancement skills, (5) "meaning making" (i.e. collaboratively identifying the personal significance of events), (6) identification of core patterns from dyad relationship history, (7) techniques to shift emotional responses, (8) techniques to increase emotional attunement, and (9) techniques to increase attunement to care-recipient needs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Experimental): Caregiver and patient with dementia dyads who receive the family intervention.
  Interventions: Behavioral: Telemental Health Family Intervention

INTERVENTIONS:
Behavioral: Telemental Health Family Intervention — Approximately 12-16 session family intervention that will include the following specific strategies, the implementation of which will be tailored by clinicians to the specific interpersonal deficits identified in an assessment: (1) psychoeducation on dementia, (2) communication and problem solving skills, (3) safety building skills, (4) relationship satisfaction enhancement skills, (5) "meaning making" (i.e. collaboratively identifying the personal significance of events), (6) identification of core patterns from dyad relationship history, (7) techniques to shift emotional responses, (8) techniques to increase emotional attunement, and (9) techniques to increase attunement to care-recipient needs

SUMMARY:
Dementia impacts Veterans, their families, and other Veterans who serve as caregivers. One of the most stressful aspects of caregiving is the management of behavioral problems (e.g. wandering, agitation, and sleep difficulties), which exacerbate health issues for both caregivers and persons with dementia (PWD). Existing VA caregiver treatments for caregiver stress and behavioral problems are often ineffective. Many caregivers do not realize their interactions with PWD contribute to behavioral problems and thus do not ask for help to improve their interpersonal skills. The aim of this project is to develop an assessment of interpersonal skills deficits and a related treatment strategy to assist family caregivers of PWD who are challenged by a lack of interpersonal skills and are not helped by existing family caregiver treatments. This project, will develop and test (1) a video assessment of caregiver/PWD interaction that clinicians will use to identify interpersonal difficulties and (2) a family therapy for the interpersonal difficulties clinicians identify in the assessment.

DETAILED DESCRIPTION:
Study temporarily suspended due to COVID risk associated with at risk population of Veterans with Dementia and often older caregivers.

ELIGIBILITY:
Inclusion Criteria:

Either the caregiver or the care-recipient must be a Veteran.

The caregiver must:

* Be the primary unpaid family or friend who helps or supports an individual with dementia
* Be involved in the care of the person with dementia (at least 4 hours of care per day)
* Report that the care-recipient exhibits behavioral problems that are distressing
* Not be currently receiving the REACH VA protocol

Additionally, the care-recipient must:

* Must have a documented diagnosis of dementia
* Have cognitive impairment (MMSE<23 or SLUMS<20 or diagnosis of dementia based on chart review)
* Be out of bed and able to respond to a caregiver's instructions or interventions

Exclusion Criteria:

* Caregiver severe cognitive impairment
* Caregiver inability to meet study demands
* Caregiver psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cory K. Chen, PhD, Principal Investigator — Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY
Locations (1):
- Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 dyads were enrolled
Period: Overall Study
Arm/Group | Intervention Group
Started | 4 (4 dyads were enrolled)
Caregivers | 4
Completed | 0
Not Completed | 4
Not completed — Insufficient enrollment for intervention development | 4

BASELINE CHARACTERISTICS:
Population: The Overall Number of Baseline Participants reflects individual participants, not dyads.
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants] — Population: The Overall Number of Baseline Participants reflects individual participants, not dyads.
  Participants
    Patients: number analyzed (Participants) | 4
    Patients: <=18 years | 0
    Patients: Between 18 and 65 years | 0
    Patients: >=65 years | 4
    Caregivers: number analyzed (Participants) | 4
    Caregivers: <=18 years | 0
    Caregivers: Between 18 and 65 years | 1
    Caregivers: >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] — Population: The Overall Number of Baseline Participants reflects individual participants, not dyads.
  years
    Patients: number analyzed (Participants) | 4
    Patients | 75 [55 to 87]
    Caregivers: number analyzed (Participants) | 4
    Caregivers | 69 [55 to 87]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Overall Number of Baseline Participants reflects individual participants, not dyads.
  Participants
    Patients: number analyzed (Participants) | 4
    Patients: Female | 0
    Patients: Male | 4
    Caregivers: number analyzed (Participants) | 4
    Caregivers: Female | 4
    Caregivers: Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Overall Number of Baseline Participants reflects individual participants, not dyads.
  Participants
    Patients: number analyzed (Participants) | 4
    Patients: Hispanic or Latino | 2
    Patients: Not Hispanic or Latino | 2
    Patients: Unknown or Not Reported | 0
    Caregivers: number analyzed (Participants) | 4
    Caregivers: Hispanic or Latino | 2
    Caregivers: Not Hispanic or Latino | 2
    Caregivers: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Overall Number of Baseline Participants reflects individual participants, not dyads.
  Participants
    Patients: number analyzed (Participants) | 4
    Patients: American Indian or Alaska Native | 0
    Patients: Asian | 0
    Patients: Native Hawaiian or Other Pacific Islander | 0
    Patients: Black or African American | 0
    Patients: White | 2
    Patients: More than one race | 0
    Patients: Unknown or Not Reported | 2
    Caregivers: number analyzed (Participants) | 4
    Caregivers: American Indian or Alaska Native | 0
    Caregivers: Asian | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0
    Caregivers: Black or African American | 0
    Caregivers: White | 2
    Caregivers: More than one race | 0
    Caregivers: Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Healthy Aging Brain Center Monitor (HABC Monitor):
Description: A 31-item caregiver assessment of dementia severity, caregiver stress, and mood. Contains three patient symptom domains (Cognitive, functional, behavioral/psychological) and a caregiver quality of life domain. Shown to have good internal consistency (0.73-0.92) and construct validity.
Time Frame: Post Treatment, an average of 12-18 weeks
Population: Not applicable as due to insufficient recruitment, phase I of the project was not completed and so a treatment protocol could not be developed and implemented. No data was obtained as the intervention phase of the study did not begin.
Arm/Group | Intervention Group
Number analyzed (Participants) | 0

2. Secondary Outcome: The Kansas Marital Conflict Scale (KMCS)
Description: A 37-item self-report scale consisting of three subscales of how well partners are able to: (1) listen and understand each other's perspectives, (2) express his or her point of view , and (3) come to a mutually satisfactory compromise. It has been shown to have high internal consistency ( = .87 to .90) and test-retest reliability (r = .62 to .92). Although developed for marital relationships, all items are applicable or easily modified for a variety of interpersonal relationships.
Time Frame: Post Treatment, an average of 12-18 weeks
Population: as for outcome 1
Arm/Group | Intervention Group
Number analyzed (Participants) | 0

3. Secondary Outcome: Patient Health Questionnaire - 9 (PHQ)
Description: A 9-item self-report scale based on DSM-IV criteria for Major Depressive Disorder, has been shown to have good sensitivity and specificity and is predictive of health outcomes such as sick days, clinic visits, and symptom related difficulty. Internal reliability of the PHQ-9 is excellent ( = 0.89).
Time Frame: Post Treatment, an average of 12-18 weeks
Population: as for outcome 1
Arm/Group | Intervention Group
Number analyzed (Participants) | 0

4. Secondary Outcome: Zarit Burden Scale
Description: A 12-item self-report scale shown to have acceptable indices of internal consistency for the two distinct factors of the scale - personal strain and role strain ( =0.88 and =0.78) and a good predictor of caregiver mental health outcomes.
Time Frame: Post Treatment, an average of 12-18 weeks
Population: as for outcome 1
Arm/Group | Intervention Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Not applicable as the intervention was ultimately not provided given the lack of sufficient initial recruitment during phase I of the project which involved development of the intervention.
Description: Not collected as the study did not progress to a phase where the intervention was delivered and so no adverse events were relevant to the sample (as no intervention was delivered).
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03116464/Prot_SAP_000.pdf